CLINICAL TRIAL: NCT03187574
Title: A Prospective Comparison of Two Vaginal Mesh Kits in the Management of Anterior and Apical Vaginal Prolapse: Long Term-results for Apical Fixation and Quality of Life
Brief Title: Comparison of Two Vaginal Mesh Kits in the Management of Vaginal Prolapse
Acronym: ELEPE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0356
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Vaginal Prolapse
Keywords: vaginal prolapse, mesh kit, anatomic assessment, quality of life
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: group received Elevate Ant™ single-incision mesh
  Interventions: Device: Elevate Ant™
- Group B: group received Perigee™ transvaginal mesh
  Interventions: Device: Perigee™

INTERVENTIONS:
Device: Elevate Ant™ — Surgery with Elevate Ant™
  Groups: Group A
Device: Perigee™ — Surgery with Perigee™
  Groups: Group B

SUMMARY:
Our study is a non-randomized prospective study compared two groups matched for anterior/apical POP-Q grade: 84 received Elevate Ant™ single-incision mesh (group A) and 42 Perigee™ transvaginal mesh (group B). The study hypothesis was that the Elevate Ant™ mesh would provide better apical correction than the Perigee™ mesh. One- and 2-year follow-up comprised anatomic assessment (POP-Q) and QoL (PFDI-20, PFIQ-7, PISQ-12). Success was defined as 2-year POP-Q ≤1. Secondary endpoints were function and complications.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patient presenting with POP-Q grade ≥3 anterior or apical prolapse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with grade ≥3 anterior prolapse
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
comparison of anatomic correction rates in the vaginal apex at 1 year between two mesh kits | 1 year post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gery LAMBLIN, Principal Investigator — Hospices Civils de Lyon

IPD SHARING:
Plan to Share IPD: No